CLINICAL TRIAL: NCT05707819
Title: Sintilimab (PD-1 Antibody) in Combination With Chemoradiotherapy in High-risk Locoregionally-advanced Nasopharyngeal Carcinoma: a Single-arm, Multicentre, Phase 2 Trial
Brief Title: Sintilimab in Combination With Chemoradiotherapy in High-risk Locoregionally-advanced Nasopharyngeal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, Principal Investigator, Cancer Hospital of Guangxi Medical University
Other Study IDs: CS2021(124)
Record Dates: First submitted 2022-07-29; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Nasopharyngeal Carcinoma; Sintilimab
Keywords: Nasopharyngeal Carcinoma; Sintilimab; high risk
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — sintilimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sintilimab+Chemoradiotherapy: Patients will receive 3 cycles of induction chemotherapy with gemcitabine and cisplatin and concurrent cisplatin-radiation plus Sintilimab, and then receive 11 cycles of Sintilimab after intensity-modulated radiotherapy (IMRT). All patients will receive IMRT. Sintilimab will begin on day 1 of induction chemotherapy and continue every 3 weeks for 17 cycles.
  Interventions: Drug: Sintilimab (PD-1 Antibody)

INTERVENTIONS:
Drug: Sintilimab (PD-1 Antibody) — Patients will receive 3 cycles of induction chemotherapy with gemcitabine and cisplatin and concurrent cisplatin-radiation plus Sintilimab, and then receive 11 cycles of Sintilimab after intensity-modulated radiotherapy (IMRT). All patients will receive IMRT. Sintilimab will begin on day 1 of induction chemotherapy and continue every 3 weeks for 17 cycles.
  Other Names: PD-1

SUMMARY:
The program aims to enroll patients with stage high risk (AJCC 8th, T3-4N2-3M0) . Patients will receive 3 cycles of induction chemotherapy with gemcitabine and cisplatin and concurrent cisplatin-radiation plus Sintilimab, and then receive 11 cycles of Sintilimab after intensity-modulated radiotherapy (IMRT). All patients will receive IMRT. Sintilimab will begin on day 1 of induction chemotherapy and continue every 3 weeks for 17 cycles.

DETAILED DESCRIPTION:
The program aims to enroll patients with stage high risk (AJCC 8th, T3-4N2-3M0) locoregionally advanced nasopharyngeal carcinoma (LANPC). Patients will receive 3 cycles of induction chemotherapy with gemcitabine and cisplatin and concurrent cisplatin-radiation plus Sintilimab (200mg q3wk), and then receive 11 cycles of Sintilimab after intensity-modulated radiotherapy (IMRT). All patients will receive IMRT. IMRT：PGTVnx: 69.96 Gy /33f, PGTVnd: 66~70 Gy /33f, PCTVnd: 63~64 Gy/33f, PCTV1: 60~62 Gy/33f, PCTV2: 54~56 Gy/33f. Sintilimab will begin on day 1 of induction chemotherapy and continue every 3 weeks for 17 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed Non-keratinizing nasopharyngeal carcinoma.
2. Tumor staged as III-IVA (AJCC 8th, T3-4N2-3M0).
3. Eastern Cooperative Oncology Group performance status ≤1.
4. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.
5. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.
6. Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
7. Patients must be informed of the investigational nature of this study and give written informed consent.
8. Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug.

Exclusion Criteria:

* 1.Age > 70 or < 18. 2.Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA >1×10e3 copies/ml or 200IU/ml 3.Hepatitis C virus (HCV) antibody positive 4.Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment.

  5.Has a known history of interstitial lung disease. 6.Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroid will be allowed.

  7.Has received a live vaccine within 30 days before informed consent or will receive a live vaccine in the near future.

  8.Is pregnant or breastfeeding. 9.Has a history of other malignancies except carcinoma in situ, adequately treated non-melanoma skin cancer, and papillary thyroid cancer.

  10.Has known allergy to large molecule protein products or any compound of sintilimab.

  11.Has a known history of human immunodeficiency virus (HIV) infection. 12.Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk Locoregionally-advanced nasopharyngeal carcinoma
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 5 years
  Defined from date of recruit to date of first documentation of progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Defined from date of recruit to date of first documentation of death from any cause or censored at the date of the last follow-up.
Locoregional Relapse-Free Survival (LRRFS) | 5 years
  Defined from date of recruit to date of first documentation of locoregional relapse or until the date of the last follow-up visit.
Distant Metastasis-Free Survival (DMFS) | 5 years
  Defined from date of recruit to date of first documentation of distant metastases or until the date of the last followup visit.
Objective Response Rate （ORR） | through study completion, an average of 1 year
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using RECIST v1.1Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI).
Incidence rate of adverse events (AEs) | 5 years
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
Serious adverse events (SAE) | 5 years
  Serious adverse events (SAE) is defined as either death, life-threatening, or Permanent or severe disability/incapacity.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Dong Zhu, Doctor, Principal Investigator — Cancer Hospital of Guangxi Medical University; Ling Li, Master, Principal Investigator — Cancer Hospital of Guangxi Medical University
Locations (1):
- Guangxi Medical University Cancer Hospital, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No